CLINICAL TRIAL: NCT06792877
Title: Mechanisms of Mindfulness for Cognition in Early-Stage Alzheimer's Disease
Brief Title: Mindfulness for Cognition in Early-stage Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Turk, Behavioral Neurologist at VA Boston Memory Disorders Clinic; Assistant Professor of Neurology at Boston University Chobanian & Avedisian School of Medicine, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1796795
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease; TBI (Traumatic Brain Injury); Aging; Healthy Elderly; Alzheimer&Amp;Amp;#39;s Dementia (AD)
Keywords: Mindfulness; Aging; Mild Cognitive Impairment (MCI); Cognition; Memory; Alzheimers Disease; Social Group
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries, Traumatic; Alzheimer Disease | interventions — Mindfulness-Based Stress Reduction; Meditation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness (Experimental): MBSR course of mindfulness using focused attention, body scan practice and light chair yoga.
  Interventions: Behavioral: Mindfulness Intervention; Behavioral: Waitlist then mindfulness
- Mindfulness Waitlist (No Intervention): Individuals in the Mindfulness Waitlist group will not engage in any of the study interventions until 2 months has passed. Then they will be enrolled in the Mindfulness Intervention.

INTERVENTIONS:
Behavioral: Mindfulness Intervention — The Mindfulness Intervention is an adapted form of Mindfulness-based stress reduction (MBSR) training virtual class that meets for 10 weeks. The class involves mindfulness training using awareness and focused attention, group discussion of the experience, and mindful movement. The Mindfulness Intervention also includes daily home practice using mindfulness recordings.
  Other Names: Mindfulness-Based Stress Reduction; Meditation
  Arms: Mindfulness
Behavioral: Waitlist then mindfulness — Participants in this arm will first wait 10 weeks and then complete a mindfulness course with outcome measures assessed at baseline, after 10 weeks wait list and then after mindfulness course.
  Arms: Mindfulness

SUMMARY:
The goal of this clinical trial is to learn if mindfulness meditation can improve outcomes in older adults with and without cognitive impairment. The main questions it aims to answer are:

1. How does mindfulness impact thinking and memory?
2. How does mindfulness influence brain function and structure?
3. How does mindfulness affect daily function and quality of life?

Researchers will compare all outcomes to one other groups. In one group, individuals will participate in a mindfulness class intervention; in the other group, individuals will not engage in any active interventions immediately, but will be placed on a waitlist for the mindfulness intervention. Researchers will compare all outcomes between the groups groups to determine whether the mindfulness interventions leads to greater improvement compared to no intervention (waitlist group).

Participants will:

* Be randomly assigned to participate in the mindfulness intervention, or no immediate intervention (waitlist)
* Complete paper-and-pencil cognitive testing, surveys, computerized tasks, and neuroimaging measures (EEG and MRI) before and after the intervention

Outcomes will be assess at baseline, 2 months, 4 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older adults will show cognitive performance within 1.0 SD for age & education adjusted norms on a neuropsychological test battery
* Mild cognitive impairment (MCI) participants will show performance on delayed recall or one more or more other cognitive domains worse than 1.5 SD for age & education adjusted norms, an MMSE score between 25-30, and a MoCA score between 20-30.

Exclusion Criteria:

* Participants without a computer, smart phone and internet access will be excluded
* If they cannot understand the informed consent form or have moderate dementia.
* Mood disorders (e.g., PTSD, depression, anxiety) or alcohol and drug use that either interferes with day-to-day life or required hospitalization within the past 5 years
* Cerebrovascular disease
* Any medical condition whose severity could significantly impair cognition (e.g., stroke, frontotermporal dementia, Parkinson's disease) are exclusionary

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological tests | From before the intervention (baseline) to after the intervention (post-intervention 10 weeks)
  Paper-and-pencil tests measuring attention, processing speed, and memory.
Performance on computerized tasks | From before the intervention (baseline) to after the intervention (post-intervention 10 weeks)
  Reaction time and accuracy on computer tasks measuring attention and memory
Resting state and event-related electrophysiology | From before the intervention (baseline) to after the intervention (post-intervention 10 weeks)
  Electrophysiology measured while at rest and time-locked to performance on a computerized task measuring attention and memory
Brain function and structure | From before the intervention (baseline) to after the intervention (post-intervention 10 weeks))
  Blood-oxygen-level-dependent (BOLD) for functional magnetic resonance imaging. Voxel-based morphometry (VBM) and diffusion tensor imaging (DTI) for structural magnetic resonance imaging.
Survey outcomes | From before the intervention (baseline) to after the intervention (post-intervention 10 weeks))
  Surveys measuring mood, social isolation, sleep, and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- VA Boston Healthcare System - Jamaica Plain Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided